CLINICAL TRIAL: NCT02492789
Title: An Open-Label, Multicenter, Nonrandomized, Dose-Escalation and Tumor-Expansion Phase 1 Study to Evaluate the Safety and Tolerability of INCSHR01210 (Formerly SHR-1210) in Subjects With Advanced Solid Tumors
Brief Title: A Trial to Evaluate Safety and Tolerability of INCSHR01210 in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCSHR1210-101
Record Dates: First submitted 2015-06-26; First posted 2015-07-09 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumors and Hematologic Malignancy
Keywords: immunotherapy; solid tumor; PD-1 blockade
MeSH Terms: conditions — Hematologic Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INCSHR01210 (Experimental): 3 dose levels are designed in this study.3 to 6 patients (traditional "3+3" design) will be enrolled in each dose cohort. INCSHR01210 injection at each dose level is administered every 2 weeks (q2w, except in the first cycle).
  Interventions: Biological: INCSHR01210 injection

INTERVENTIONS:
Biological: INCSHR01210 injection — Part1: INCSHR01210 injection at a dose of 1, 3 or 10 mg/kg is administered every 2 weeks (3+3,q2w, except in the first cycle, in which subjects will be only dosed once on Day 1 for PK samplings and dose limiting toxicity observation). Response is assessed by every 2 cycles (4 weeks each cycle) by using irRECIST.
  Part2: Additional patients (200mg dose cohorts will be enrolled in Part 2, depending on the data outcomes in Part 1, to further explore preliminarily clinical benefits of INCSHR01210 as well as the other objectives of the study.
  Other Names: SHR-1210; HR-301210

SUMMARY:
This is an open-label, multicenter, non-randomized, dose escalation and tumor-expansion phase I trial to evaluate safety and tolerability of INCSHR01210 in patients with advanced solid tumors. The trial will enroll subjects with advanced solid tumor who have failed current standard anti-tumor therapies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age;
* Patients diagnosed with solid tumors histologically or cytologically and documented as advanced or metastatic disease for which there is no known effective anti-tumour treatment (refractory to or relapsed from standard therapies);
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
* Life expectancy ≥ 12 weeks;
* Patients enrolled to Part 2 Expansion Cohorts:

  * must have measurable lesion(s) according to the RECIST v1.1;
  * Cohort A (endometrial carcinoma): Subjects diagnosed with histologically confirmed advanced or metastatic endometrial carcinoma (sarcomas and mesenchymal tumors are excluded). Subjects must have relapsed or be refractory to at least 1 prior standard therapy in the metastatic setting, have been intolerant to standard therapies, or have refused standard therapy. In addition, subjects with disease recurrence within 12 months of completion of adjuvant therapy are eligible.
  * Cohort B (thymic carcinoma): Subjects diagnosed with histologically or cytologically confirmed advanced or metastatic thymic carcinoma based on local guidelines.
  * Cohort C (biliary tract carcinoma): Subjects diagnosed with histologically or cytologically confirmed, advanced or metastatic extrahepatic cholangiocarcinoma (carcinoma of the gallbladder or biliary tree) or carcinoma of the ampulla of Vater. Subjects must have relapsed or be refractory to at least 1 prior standard therapy, have been intolerant to standard therapies, or have refused standard therapy.
  * Cohort D (CUP): Subjects diagnosed with CUP based on ESMO guidelines.
* Adequate laboratory parameters at screening period as evidenced by:

  * Absolute neutrophil count ≥ 1.5×109/L (1,500/mm3)
  * Platelets ≥100×109/L (100,000/mm3)
  * Hemoglobin ≥ 9.0 g/dL (90 g/L)
  * Albumin levels ≥ 2.8 g/dL
  * Total bilirubin ≤ 1.5×ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN; for patients with liver metastases, ALT and AST ≤ 5×ULNSerum creatinine ≤ 1.5×ULNAble to understand and sign an informed consent.

Exclusion Criteria:

Subjects who fulfill any of the following criteria at screening will be ineligible for admission:

* Subjects with any active autoimmune disease or history of autoimmune disease, or history of syndrome that requires systemic steroids or immunosuppressive medications, including but not limited to the following: rheumatoid arthritis, pneumonitis, colitis (inflammatory bowel disease), hepatitis, hypophysitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Subjects with the following conditions will not be excluded from this study: asthma that requires intermittent use of bronchodilators, hypothyroidism stable on hormone replacement, vitiligo, Graves' disease, or Hashimoto's disease. Additional exceptions may be made with medical monitor approval.
* Known history of hypersensitivity to any components of the INCSHR01210 formulation.
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration. Note: corticosteroids used for the purpose of intravenous contrast allergy prophylaxis are allowed.
* Active CNS metastases (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive disease). Subjects with brain or meningeal metastases that were previously treated must be clinically stable (magnetic resonance imaging at least 4 weeks apart do not show evidence of new or enlarging metastases) and have discontinued immunosuppressive doses of systemic steroids (> 10 mg/day prednisone or equivalent) for at least 2 weeks before study drug administration.
* Uncontrolled clinically significant medical condition, including but not limited to the following: (1) congestive heart failure (New York Health Authority Class > 2), (2) unstable angina, (3) myocardial infarction within the past 12 months, or (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention.
* Prior systemic chemotherapy (< 6 weeks if chemotherapy including nitrosoureas or mitomycin), radiotherapy, immunotherapy, hormone therapy, surgery or target therapy within 4 weeks before the study drug administration, or any unresolved adverse events > CTCAE Grade 1 (with the exception of any stable chronic toxicities not expected to resolve).
* Active infection or an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, subjects with tumor fever may be enrolled).
* History of immunodeficiency including seropositivity for human immunodeficiency virus, or other acquired or congenital immune-deficient disease.
* Any other medical (eg, pulmonary, metabolic, congenital, endocrinal or CNS disease), psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.
* Investigational therapy administered within 4 weeks before the first dose of INCSHR01210.
* Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation based on institutional guidelines and tests. Testing may include the following: HBV DNA, HCV RNA, hepatitis B surface antigen, or anti-hepatitis B core antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2015-09-01; Primary Completion 2019-03-01 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 15 months
  Recommended phase II doses (RP2D) is 200 mg, and the only dose interval to be tested will be once every 4 weeks (Q4W).

SECONDARY OUTCOMES:
Pharmacokinetics (PK) profile of INCSHR01210 (Tmax) | Day 1 of cycle 1
Maximum tolerated dose (MTD) of INCSHR01210 | 6 months
Incidence of anti-INCSHR01210 antibody in serum | 15 months
PD-1 receptor occupancy | 15 months
Duration of response | 15 months
Objective response rate | 15 months
Time to progression | 15 months
Pharmacokinetics (PK) profile of INCSHR01210 (Cmax) | Day 1 of cycle 1
Pharmacokinetics (PK) profile of INCSHR01210 (AUC0-28day) | Day 28 of cycle 1
Pharmacokinetics (PK) profile of INCSHR01210 (accumulation ratio R) | Day 28 of each cycle

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Austin Hospital/Olivia Newton-John Cancer Research Institute, Heidelberg, Victoria
  - Blacktown Hospital, Blacktown
  - Chris O'Brien Life House, Camperdown
  - Nucleus Network, Melbourne
  - Linear Clinical Research Limited, Nedlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lickliter JD, Gan HK, Voskoboynik M, Arulananda S, Gao B, Nagrial A, Grimison P, Harrison M, Zou J, Zhang L, Luo S, Lahn M, Kallender H, Mannucci A, Somma C, Woods K, Behren A, Fernandez-Penas P, Millward M, Meniawy T. A First-in-Human Dose Finding Study of Camrelizumab in Patients with Advanced or Metastatic Cancer in Australia. Drug Des Devel Ther. 2020 Mar 18;14:1177-1189. doi: 10.2147/DDDT.S243787. eCollection 2020. PMID 32256049